CLINICAL TRIAL: NCT01485432
Title: Can Goal Directed Hemodynamic Management Improve Renal Outcome After Renal Transplant Surgery?
Brief Title: Goal Directed Hemodynamic Management and Renal Outcome After Renal Transplant Surgery
Acronym: IROR
Status: Terminated | Type: Observational
Why Stopped: Low recruitment of patients.
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: IROR
Record Dates: First submitted 2011-11-11; First posted 2011-12-05 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Renal Transplant Surgery
Keywords: Renal transplant surgery; hemodynamic management; PiCCO; delayed graft function
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- P group: Group P: Fluid Management according to measurements with PiCCO®
  Interventions: Device: PiCCO® Monitoring
- C group: Group C: Conventional fluid management

INTERVENTIONS:
Device: PiCCO® Monitoring — Fluid and vasopressor management according to PiCCO measurements
  Groups: P group

SUMMARY:
This study is designed to compare the incidence of delayed graft function in patients following renal transplant surgery with different perioperative hemodynamic managements: a goal directed hemodynamic management group (using PiCCO) and a control group.

DETAILED DESCRIPTION:
Volume assessment and management during renal transplantation is one of the most challenging problems the anesthetist has to deal with. It seems sensible that individualized volume management and hydration therapy during the operation and during the stay at the intensive care unit could improve perfusion of the transplanted organ resulting in a better transplant function. Aim of this study is to investigate the impact of a goal directed hemodynamic management on incidence of delayed graft function (DGF) after renal transplant surgery.

Therefore patients will be randomized in one of two groups, the PiCCO group with goal directed hemodynamic management during operation and during the ICU-stay and the control group with hemodynamic management performed according to heart rate, blood pressure and central venous pressure.

ELIGIBILITY:
Inclusion Criteria:

* Renal Transplant Surgery
* Age ≥ 65 years
* Written informed consent

Exclusion Criteria:

* Contraindications for an arterial line in the femoral artery:

  * stents
  * bypasses
  * severe peripheral artery occlusive disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing renal transplant surgery
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
delayed graft function | Start of anesthesia until day 7 after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Jungwirth, MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Ismaninger Str. 22, 81675 München
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Goepfert MS, Reuter DA, Akyol D, Lamm P, Kilger E, Goetz AE. Goal-directed fluid management reduces vasopressor and catecholamine use in cardiac surgery patients. Intensive Care Med. 2007 Jan;33(1):96-103. doi: 10.1007/s00134-006-0404-2. Epub 2006 Nov 21. PMID 17119923
- [Background] Boom H, Mallat MJ, de Fijter JW, Zwinderman AH, Paul LC. Delayed graft function influences renal function, but not survival. Kidney Int. 2000 Aug;58(2):859-66. doi: 10.1046/j.1523-1755.2000.00235.x. PMID 10916111